CLINICAL TRIAL: NCT05360082
Title: Direct Quantitative Comparison Between [11C]UCB-J and [18F]SynVest-1 PET as Markers for Synaptic Density in Huntington's Disease.
Brief Title: Comparison Between [11C]UCB-J and [18F]SynVest-1 PET in HD.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: CHDI Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S66610
Record Dates: First submitted 2022-04-28; First posted 2022-05-04 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2024-12

CONDITIONS: Huntington Disease
Keywords: PET; SV2A; Huntington disease; synaptic density
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 + 2: healthy controls (Active Comparator): Age -and sex matched to HD patients (to stage 3 HD patients for cohort 1 and to stage 2 HD patients for cohort 2)
  Interventions: Other: [11C]UCB-J PET; Other: [18F]SynVest-1 PET
- Cohort 1: stage 3 manifest HD patients (Experimental): * HTT CAG repeat expansion 40 - 50;
  * stage 3 as determined by the HD-ISS staging criteria;
  * UHDRS TFC >/= 10.
  Interventions: Other: [11C]UCB-J PET; Other: [18F]SynVest-1 PET
- Cohort 2: stage 2 manifest HD patients (Experimental): * HTT CAG repeat expansion 40 - 50;
  * stage 2 as determined by the HD-ISS criteria;
  * PIN score 0.47 to 1.84.
  Interventions: Other: [11C]UCB-J PET; Other: [18F]SynVest-1 PET

INTERVENTIONS:
Other: [11C]UCB-J PET — 11C-labeled SV2A binding PET radioligand
Other: [18F]SynVest-1 PET — 18F-labeled SV2A binding PET radioligand

SUMMARY:
Positron Emission Tomography (PET) is a functional imaging technique, which enables in vivo visualization of biological molecules expressed in human tissues. Brain PET is most powerful to study a vast range of neurological and psychiatric disorders in vivo, targeting neuronal and glial activity, metabolism, cerebral blood flow, receptor proteins or misfolded proteins.

In vivo imaging of synaptic density in the human brain has become feasible through development of [11C]UCB-J, a PET radioligand for the synaptic vesicle protein SV2A, which is ubiquitously and homogeneously present in presynaptic terminals throughout the brain. A first study in Huntington's disease (HD) mutation carriers showed loss of striatal [11C]UCB-J binding (also when corrected for atrophy), as well as in the neocortex (Delva et al, Neurology 2022). Moreover, regional synaptic loss was highly correlated to motor impairment.

In order to be able to use SV2A PET as widespread available biomarker tool to assess synaptic integrity, disease progression and/or response to mHTT lowering drugs, the short half-life of 11C (20 minutes) for [11C]UCB-J remains a hurdle. Recently, [18F]SynVesT-1, an optimized 18F-labeled analogue of [11C]UCB-J with similar kinetics, binding affinity, and test-retest precision properties has been evaluated in humans.

However, there is evidence from preclinical studies conducted at University of Antwerp that in the zQ175DN knock-in mouse model of HD, larger variability and lower effect-sizes are seen with [18F]SynVest-1 than with [11C]UCB-J.

In order to ascertain a similar effect size and quantification properties for [18F]SynVest-1 and [11C]UCB-J PET in human HD patients and to validate simplified measures (such as SUVR with white matter as reference region) and SynVest, this head-to-head fully quantitative study is performed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy controls (n = 10-20)

   * Subject is judged to be in good health by the investigator on the basis of medical history, physical examination including vital signs, clinical laboratory test and urinalysis.
   * No history or evidence of current major neurological, internal or psychiatric disorder, based on the medical assessment as described hereabove and neuropsychological assessment.
   * In subjects < 60 years of age, an unremarkable structural MRI scan as assessed by expert radiologist. In subjects >= 60 years of age white matter hyperintensities corresponding to a white matter lesion (WML) Fazekas score < 2 on the Age-Related White Matter changes scale are acceptable.
2. HD-ISS stage 3 HD mutation carriers (n = 10)

   * HTT CAG repeat expansion 40 - 50
   * stage 3 as determined by the HD-ISS staging criteria
   * UHDRS TFC >/= 10
3. HD-ISS stage 2 HD mutation carriers (n = 10)

   * HTT CAG repeat expansion 40 - 50
   * stage 2 as determined by the HD-ISS staging criteria
   * PIN score 0.47 - 1.84

Exclusion Criteria:

* Neuropsychiatric diseases; for HD mutation carriers any neuropsychiatric diseases other than HD
* Major internal medical diseases
* White matter lesion load on FLAIR Fazekas score 2 or higher or other relevant MRI abnormalities
* History of alcohol abuse or current alcohol abuse (chronic use of more than 15 units per week) or drug use
* Contraindications for MR
* Subject suffers from claustrophobia or cannot tolerate confinement during PET-MRI scanning procedures; subject cannot lie still for 30 minutes inside the scanner.
* Subject is unwilling to avoid unusual, unaccustomed, or strenuous physical activity (i.e., weightlifting, running, bicycling) from the time of the pre-study visit until the end of scanning.
* Subject does not understand the study procedures or does not have a guardian who understands the study procedures.
* Subject (or guardian) is unwilling or unable to perform all of the study procedures or is considered unsuitable in any way by the principal investigator.
* Subject is on anticoagulant therapy.
* Subject is pregnant (according to Ulti Med hCG urine test) or breastfeeding.
* Subject is a woman of childbearing potential who does not agree to apply appropriate contraception methods during study participation and continues to do so for at least 6 months after study completion.
* Subject is a man with a pregnant or non-pregnant WOCBP partner, who does not agree to use a condom and continue to do so until 90 days after study completion. In addition, the non-pregnant WOCBP partner should use a highly effective method of contraception.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Compare Vt of [11C]UCB-J and [18F]SynVest-1 in manifest HD and healthy controls | A first data analysis will be done when all cohort 1 subjects have undergone evaluations. A go-no-go decision will then be made before proceeding with cohort 2. Data analysis of cohort 2 subjects will follow completion of cohort 2.
  Assess whether changes in total volume of distribution (Vt) are similar for [11C]UCB-J and [18F]SynVest-1 in manifest HD compared to healthy controls.

SECONDARY OUTCOMES:
Compare variance in Vt within groups for [11C]UCB-J and [18F]SynVest-1 | A first data analysis will be done when all cohort 1 subjects have undergone evaluations. A go-no-go decision will then be made before proceeding with cohort 2. Data analysis of cohort 2 subjects will follow completion of cohort 2.
  Compare the variance in total volume of distribution (Vt) between [11C]UCB-J and [18F]SynVest-1 in healthy volunteers and manifest HD patients.
Compare simplified measures (BPND, SUVR) to assess group differences for [11]C-UCB-J and [18]F-SynVest-1 | A first data analysis will be done when all cohort 1 subjects have undergone evaluations. A go-no-go decision will then be made before proceeding with cohort 2. Data analysis of cohort 2 subjects will follow completion of cohort 2.
  Compare volume of distribution (Vt), BPND and SUVR between [11C]UCB-J and [18F]SynVest-1 in HD patients and healthy controls.

CONTACTS AND LOCATIONS:
Overall Officials: Koen Van Laere, MD, PhD, DSc, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
To be determined

REFERENCES:
- [Background] Delva A, Michiels L, Koole M, Van Laere K, Vandenberghe W. Synaptic Damage and Its Clinical Correlates in People With Early Huntington Disease: A PET Study. Neurology. 2022 Jan 4;98(1):e83-e94. doi: 10.1212/WNL.0000000000012969. Epub 2021 Oct 18. PMID 34663644
- [Background] Finnema SJ, Nabulsi NB, Eid T, Detyniecki K, Lin SF, Chen MK, Dhaher R, Matuskey D, Baum E, Holden D, Spencer DD, Mercier J, Hannestad J, Huang Y, Carson RE. Imaging synaptic density in the living human brain. Sci Transl Med. 2016 Jul 20;8(348):348ra96. doi: 10.1126/scitranslmed.aaf6667. PMID 27440727
- [Background] Naganawa M, Li S, Nabulsi N, Henry S, Zheng MQ, Pracitto R, Cai Z, Gao H, Kapinos M, Labaree D, Matuskey D, Huang Y, Carson RE. First-in-Human Evaluation of 18F-SynVesT-1, a Radioligand for PET Imaging of Synaptic Vesicle Glycoprotein 2A. J Nucl Med. 2021 Apr;62(4):561-567. doi: 10.2967/jnumed.120.249144. Epub 2020 Aug 28. PMID 32859701
- See also: CHDI Foundation, Inc. — https://chdifoundation.org/